CLINICAL TRIAL: NCT00099450
Title: Single-Center, Open-Labeled Dose Escalation Followed by Randomized, Double-Blind, Placebo-Controlled Cohort Study of the Tolerability, Pharmacokinetics, and Pharmacodynamics of INS50589 Intravenous Infusion in Healthy Volunteers
Brief Title: Study of the Tolerability, Pharmacokinetics, and Pharmacodynamics of INS50589 Intravenous Infusion in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 025-101
Record Dates: First submitted 2004-12-14; First posted 2004-12-15 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Cardiovascular Disease
Keywords: bleeding; blood transfusion; surgeries
MeSH Terms: conditions — Cardiovascular Diseases; Hemorrhage

INTERVENTIONS:
Drug: INS50589 Intravenous Infusion

SUMMARY:
The objectives of this study are to look at the safety and tolerability of the experimental drug, how people process the drug, how the drug affects people, and to identify a dose or doses to study in subsequent future studies.

DETAILED DESCRIPTION:
The purposes of this trial are to determine if administration of INS50589 Intravenous Infusion is well tolerated, to determine the pharmacological effects of INS50589 at different doses, and to identify an appropriate dose for later efficacy studies. More specifically, the objectives are to:

* Evaluate safety and tolerability
* Evaluate pharmacokinetics of INS50589 and its major metabolite(s)
* Evaluate effects of INS50589 on platelet function at various dose levels
* Evaluate potential relationship between plasma concentrations of INS50589 and various pharmacodynamic endpoints
* Identify one or more dose levels of INS50589 for future studies

ELIGIBILITY:
Inclusion Criteria:

* Have body mass index (BMI) between 18.5 kg/m2 and 35 kg/m2 and body weight no greater than 120 kg.
* If female, must not be pregnant or lactating, and if of childbearing potential or sexually active, must use acceptable method of birth control.

Exclusion Criteria:

* Have clinically significant acute or chronic disease (e.g., coronary artery disease, diabetes, chronic renal insufficiency, asthma).
* Have major surgery within eight weeks of dosing.
* Have overt viral illness within four weeks of dosing.
* Have tendency or history in family of tendency for bleeding.
* Have clinically significant abnormalities on clinical laboratory tests (chemistry, hematology, urinalysis).
* Have taken aspirin or any other non-steroidal anti-inflammatory drug (NSAID) within 10 days prior to admission to study facility.
* Have ever taken or received any of the following for medical conditions: (antiplatelet compounds including clopidogrel, ticlopidine, dipyridamole, tirofiban, eptifibatide, abciximab, adenosine, and prostacyclin) or (anticoagulants including vitamin K antagonists, thrombin inhibitors, heparins, hirudin or related compounds, argatroban and factor Xa inhibitors)
* Have a clinically significant ECG abnormality.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2004-12; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Platelet function

SECONDARY OUTCOMES:
Pilot study - not specified

CONTACTS AND LOCATIONS:
Overall Officials: Amy Schaberg, BSN, Study Director
Locations (1):
- Quintiles Phase I Services, Lenexa, Kansas, United States

REFERENCES:
- [Result] Johnson FL, Boyer JL, Leese PT, Crean C, Krishnamoorthy R, Durham T, Fox AW, Kellerman DJ. Rapid and reversible modulation of platelet function in man by a novel P2Y(12) ADP-receptor antagonist, INS50589. Platelets. 2007 Aug;18(5):346-56. doi: 10.1080/09537100701268741. PMID 17654304